CLINICAL TRIAL: NCT07040761
Title: Evaluation of Medical Literacy in Patients Who Presented With a TIA Treated in Emergency Departments in Lyon
Brief Title: Medical Literacy in TIA (Transient Ischemic Attack) Patients
Acronym: LitterAIT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0091; 2025-A00239-40 (Other: ID-RCB)
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Transient Ischemic Attack
Keywords: Transient ischemic attack; Medical literacy; Emergency department
MeSH Terms: conditions — Ischemic Attack, Transient; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIA: TIA patients diagnosed in the emergency department and sent to neurology day hospital for evaluation
  Interventions: Other: Two medical questionnaires

INTERVENTIONS:
Other: Two medical questionnaires — Medical questionnaires delivered by hand and completed the same day

SUMMARY:
There are around 30,000 TIAs (transient ischemic attacks) per year in France. This pathology can be the warning sign of a stroke, responsible for significant morbidity and mortality at the population level.

An important part of patient care is to teach them to recognize the symptoms suggestive of a stroke as well as the contributing factors, thus improving the medical literacy of patients.

The results of studies that have assessed medical literacy in France and Europe converge towards a rather low level.

Some studies have focused on stroke literacy in France. They show good knowledge of risk factors and the attitude to adopt in the event of a stroke, but recognition of symptoms remains problematic.

There is very little literature concerning knowledge of TIA in the general population and there are no studies concerning literacy in a population having presented with TIA.

The aim of this study is to evaluate the knowledge of patients who have presented with a TIA (and therefore at high cardiovascular risk) about this disease (risk factors, symptoms, severity, attitude to adopt in the event of symptoms), after their visit to the emergency room.

The investigators make the hypothesis that knowledge of TIA and its consequences will be rather low in this population of patient, even after a medical contact at the emergency room.

ELIGIBILITY:
Inclusion Criteria :

* Adult men and women ≥18 years old
* Patient referred to neurology day hospital at the Pierre Wertheimer neurological hospital after first care in the emergency department
* Patient having been informed and having expressed his non-opposition
* Patient affiliate to a social security scheme

Exclusion Criteria :

* Patient unable to complete the questionnaire
* History of stroke/TIA
* Patient who do not understand the French language
* Patient under legal protection, guardianship, curatorship, under judicial protection-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Lyon region who consulted an emergency department with a final diagnosis of TIA, and sent to the neurology day hospital of Pierre Wertheimer neurological hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Quality of responses to the medical literacy questionnaire specific to TIAs | Day 1 at inclusion
  The questionnaire contains 18 questions, open or closed. Each question will be analysed separately and the results will be expressed as a percentage of correct answer (in the case of a closed question mainly) or by specifying the different answers provided by the patients (in the case of an open question mainly)

CONTACTS AND LOCATIONS:
Overall Officials: Mathis Labeylie, DR, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Pierre Wertheimer hospital, Bron, France

IPD SHARING:
Plan to Share IPD: No